CLINICAL TRIAL: NCT06808152
Title: The Relation Between QTc Interval and Different Dialysate Calcium Concentarions in Hemodialysis Patients in Upper Egypt
Brief Title: QTc Interval Changes in Hemodialysis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashraf Gad Ahmed Ataia, residant doctor, Assiut University
Other Study IDs: QTc changes in HD patients
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Hemodialysis
Keywords: QTc interval; dialysate calcium concentarions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hemodialysis patients: patients on regular hemodialysis for not less than one year with age above 20 years & less than 60 . patients will be studied on two sessions of hemodialysis with different dialysate calcium concentrations, one by bicarbonate dialysate with calcium concentration 1.25 mmol/L, and bicarbonate dialysate with calcium concentration 1.5 mmol/L.

SUMMARY:
The aim of the study is to assess the correlation of QTc interval and sudden cardiac arrest in hemodialysis patients to the different dialysate calcium concentrations.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is the leading cause of death in hemodialysis. On hemodialysis, arrhythmias can occur during and shortly after receiving treatment, independent of traditional cardiovascular risk factors. Calcium, potassium, and magnesium may contribute to the development of arrhythmias during hemodialysis as these cations play a major role in development of the ventricular action potential and propagation of the electrical impulse. The optimal serum calcium range, and type of calcium measurement remains unclear, but KDOQI recommends that the dialysate calcium concentration be decreased as a means to maintain neutral or negative calcium balance and prevent vascular calcification. During hemodialysis, serum-ionized calcium varies directly with the dialysate calcium concentration, so a potential harmful effect of reducing calcium concentrations in the dialysate and serum of hemodialysis patients may lead to an increased risk of cardiac rhythm disturbances and sudden cardiac arrest (SCA). Changes in serum calcium, in turn, strongly affect the length of the QT interval so, such disparity in repolarization can be assessed by measuring the QT dispersion, that is, the variation in QT interval length, on a standard 12-lead electrocardiogram. This procedure has been shown to be a useful and reliable means of identifying patients at risk of ventricular arrhythmias. Accordingly, The present study is designed to evaluate the effect of dialysate calcium concentration on cardiac electrical stability during hemodialysis treatment by measuring the QT interval and QT dispersion before and after hemodialysis sessions, each with a different concentration of dialysate calcium.

ELIGIBILITY:
Inclusion Criteria:

* patients with End Stage Kidney Disease (ESKD) on regular hemodialysis (HD), for not less than one year with age above 20 years & less than 60.

Exclusion Criteria:

* Patients with multi- systemic diseases as SLE Patient with organ damage as heart failure, ischemic heart disease, decompensated liver disease & CVS Patients with organ transplantation Malignancy Patients above 60 years & below 20 years

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients on regular hemodialysis for not less than one year with age above 20 years & less than 60 . patients will be studied on two sessions of hemodialysis with different dialysate calcium concentrations, one by bicarbonate dialysate with calcium concentration 1.25 mmol/L, and bicarbonate dialysate with calcium concentration 1.5 mmol/L.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Q-T interval changes in hemodialysis patient | 6 weeks
  cardiac electrical stability during hemodialysis treatment

IPD SHARING:
Plan to Share IPD: Undecided